CLINICAL TRIAL: NCT03113305
Title: Changes in Ingestive Behaviour Following Gastric Bypass
Status: Completed | Type: Observational
Sponsor: University of Ulster (Other)
Collaborators: University College Dublin (Other); University of Florida (Other); Letterkenny University Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 16/WS/0056
Record Dates: First submitted 2017-04-06; First posted 2017-04-13 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Morbid Obesity
Keywords: Gastric bypass; Morbid obesity; Food choice; Ingestive behaviour; Food preference
MeSH Terms: conditions — Obesity, Morbid; Food Preferences

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — DNA, Plasma and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastric bypass patients: Patients planned to undergo Gastric bypass procedure. Patients will be assessed -1 month, 3-, 24-, 48- and 60 months post surgery.
- Healthy controls: Healthy controls with no planned weight loss/gain. Control participant assessments will be time-matched with patients.

SUMMARY:
The gastric bypass procedure is known to be one of the most successful treatments for morbid obesity and Type 2 diabetes mellitus, and has been shown to decrease appetite, energy intake, body weight and glycemia both in the short and long term. A number of reports hypothesise that these changes may be driven, at least in part, by positive shifts in food preferences following surgery. However, findings are drawn from self-reported dietary intakes which are beset with measurement bias, thus precluding definite conclusions.

The current work aims to directly observe food intake to test the hypothesis that after gastric bypass food intake changes in a manner which leads to beneficial outcomes on body weight when compared to weight stable control participants. Patients (n=32) with a planned gastric bypass procedure will be recruited from Phoenix Health (Ireland and England) and Letterkenny University Hospital (Ireland), alongside control participants (n=32) with no planned weight loss. All subjects will attend the Human Intervention Studies Unit (HISU), Ulster University on five occasions (1-month pre-surgery and 3, 12, 24 and 60 months post-surgery, with controls being time-matched). Study visits will be fully residential involving two overnight stays within the facility during which participants' 24-hour food intake will be covertly measured (7am-11pm Day 2 and breakfast Day 3) and the following procedures undertaken; basal metabolic rate, body composition, bone health, assessment of liking/wanting high fat foods and post-meal gut hormone responses. On each study visit participants will have ad lib access to a range of foods of varying macronutrient composition and which are compatible with their stated food preferences (assessed prior to the start of the study). Changes in all ingestive behaviours will be evaluated over time as compared to the control participants.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Planned gastric bypass surgery (patients only)
* No planned weight loss/gain (controls only)

Exclusion Criteria:

Patients

* Significant dysphagia, gastric outlet obstruction or any other factor which prevents consumption of a meal
* Systemic or gastrointestinal condition which may affect food intake or preference
* Pregnancy / lactation
* Significant food allergy or dietary restriction
* Medication with documented effect on food intake or food preference
* Any other physical or psychological condition which would affect the outcome of the study as determined by Phoenix Health care team.

Controls

* Medication with documented effect on food intake / preference or study outcomes
* Pregnancy / lactation
* Significant food allergy or dietary restriction
* Undertaking a weight-loss programme or planning to.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients planning to undergo gastric bypass surgery. Control participants with no planned weight loss/gain.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Food intake | Change from pre-surgery (-1 month) at 3-, 24-, 48- and 60-months post surgery
  Total energy density (kJ / gram)

SECONDARY OUTCOMES:
Total energy intake | Change from pre-surgery (-1 month) at 3-, 24-, 48- and 60-months post surgery
  24-hour intake (kJ)
Relative macronutrient intake | Change from pre-surgery (-1 month) at 3-, 24-, 48- and 60-months post surgery
  % contribution of macronutrient to energy intake
Food preferences | Change from pre-surgery (-1 month) at 3-, 24-, 48- and 60-months post surgery
  Explicit and implicit food preferences measured by the Leeds Food Preference Questionnaire
Eating occasion size | Change from pre-surgery (-1 month) at 3-, 24-, 48- and 60-months post surgery
  Grams and kJ over 24 hour period
Eating speed | Change from pre-surgery (-1 month) at 3-, 24-, 48- and 60-months post surgery
  g/min and kJ/min over 24 hour period
Meal frequency | Change from pre-surgery (-1 month) at 3-, 24-, 48- and 60-months post surgery
  Defined as a continuous period of feeding terminated with a pause >5mins
Basal Metabolic Rate | Change from pre-surgery (-1 month) at 3-, 24-, 48- and 60-months post surgery
  Measured by indirect calorimetry
Percentage body fat | Change from pre-surgery (-1 month) at 3-, 24-, 48- and 60-months post surgery
  Measured by dual X-ray absorptiometry
Percentage lean weight | Change from pre-surgery (-1 month) at 3-, 24-, 48- and 60-months post surgery
  Measured by dual X-ray absorptiometry
Bone health | Change from pre-surgery (-1 month) at 3-, 24-, 48- and 60-months post surgery
  Measured by dual X-ray absorptiometry
Serum lipid profile | Change from pre-surgery (-1 month) at 3-, 24-, 48- and 60-months post surgery
Plasma micronutrient status | Change from pre-surgery (-1 month) at 3-, 24-, 48- and 60-months post surgery
Serum C-Reactive Protein | Change from pre-surgery (-1 month) at 3-, 24-, 48- and 60-months post surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Letterkenny University Hospital, Letterkenny, Ireland
- Human Intervention Studies Unit, Ulster University, Coleraine, Co.Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Livingstone MBE, Redpath T, Naseer F, Boyd A, Martin M, Finlayson G, Miras AD, Bodnar Z, Kerrigan D, Pournaras DJ, le Roux CW, Spector AC, Price RK. Food Intake Following Gastric Bypass Surgery: Patients Eat Less but Do Not Eat Differently. J Nutr. 2022 Nov;152(11):2319-2332. doi: 10.1093/jn/nxac164. Epub 2022 Jul 23. PMID 36774099